CLINICAL TRIAL: NCT00075101
Title: Sleep, Fatigue, and Dexamethosone in Childhood Cancer
Brief Title: Sleep, Fatigue, and Dexamethosone in Children With Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Pamela S. Hinds, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NR007610-01 (NIH)
Record Dates: First submitted 2004-01-02; First posted 2004-01-05 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia
Keywords: Drug Adverse Effect; Pediatric Cancer
MeSH Terms: conditions — Leukemia; Drug-Related Side Effects and Adverse Reactions; Neoplasms | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Cycle (Experimental)
  Interventions: Drug: Dexamethosone

INTERVENTIONS:
Drug: Dexamethosone — 10 day study cycle: 5 day observation pre-steroid,5 day observation post-steroid
  Other Names: Mestinon

SUMMARY:
The purpose of this study is to determine the relationship between dexamethosone (steroid) and children's sleep and fatigue.

DETAILED DESCRIPTION:
Approximately 134 children and adolescents will be enrolled. All children and adolescents will wear a wrist actigraph for two consecutive 5-day study periods. Children and adolescents will have blood drawn 2 times on Day 1 when they are on dexamethosone. Their parents will complete a sleep diary and fatigue questionnaire by telephone on Days 2 and 5 of both study periods.

ELIGIBILITY:
Children and adolescents with Leukemia, both genders

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2000-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Fatigue and sleep quality changes | 10 days

SECONDARY OUTCOMES:
Pharmacogenetics with dextamethasone use | 5 days
Pharmacokinetics with dextamethasone use | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Hinds, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children Research Hospital, Memphis, Tennessee, United States